CLINICAL TRIAL: NCT06609486
Title: Clinical Evaluation of Bionet Sphygmomanometer Module BN1 Based on ISO 81060-2:2018 Protocol
Brief Title: Clinical Evaluation of the Performance of Bionet Sphygmomanometer Modules Based on Protocol Presented by the International Organization for Standardization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoon-Ki Park (Other)
Collaborators: Bionet Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, Hoon-Ki Park, Professor, Hanyang University Seoul Hospital
Organization: Hanyang University Seoul Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HKPark
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Blood Pressure
Keywords: Hypotension; Hypertension; Prehypertension; Sphygmomanometers
MeSH Terms: conditions — Hypotension; Hypertension; Prehypertension

STUDY DESIGN:
Intervention Model Description: In this study, the protocol applied to automatic electronic blood pressure system module BN1 for performance evaluation is ISO's proposed "ISO 81060-2:2018 Non-invasive sphygmomanometers- Part2: Clinical investment of internal automatic measurement type". The initial BP measurement is performed alternately, measuring the blood pressure by the measurer and the test device once each, and measuring blood pressure by the measurer four times by the observer and three times by the test device.
Masking Description: In this study, the protocol applied to automatic electronic blood pressure system module BN1 for performance evaluation is ISO's proposed "ISO 81060-2:2018 Non-invasive sphygmomanometers- Part2: Clinical investment of internal automatic measurement type". The initial BP measurement is performed alternately, measuring the blood pressure by the measurer and the test device once each, and measuring blood pressure by the measurer four times by the observer and three times by the test device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blood pressure measurement group (Experimental): In this study, the protocol applied to automatic electronic blood pressure system module BN1 for performance evaluation is ISO's proposed "ISO 81060-2:2018 Non-invasive sphygmomanometers- Part2: Clinical investment of internal automatic measurement type". The initial BP measurement is performed alternately, measuring the blood pressure by the measurer and the test device once each, and measuring blood pressure by the measurer four times by the observer and three times by the test device.
  Interventions: Device: Blood pressure measurement group

INTERVENTIONS:
Device: Blood pressure measurement group — In this study, the protocol applied to automatic electronic blood pressure system module BN1 for performance evaluation is ISO's proposed "ISO 81060-2:2018 Non-invasive sphygmomanometers- Part2: Clinical investment of internal automatic measurement type". The initial BP measurement is performed alternately, measuring the blood pressure by the measurer and the test device once each, and measuring blood pressure by the measurer four times by the observer and three times by the test device.

SUMMARY:
According to INTERNATIONAL STANDARD (hereafter ISO) blood pressure (BP) monitor clinical evaluation protocol (ISO 81060-2:2018, Non-invasive sphygmomanometers- Part2: Clinical investigation of intermittent automated measurement type) for BN1 (BNiBP), an electronic sphygmomanometer module newly developed by Bionet Co., Ltd., the clinical group and evaluation criteria presented in, the effectiveness of blood pressure measurement performance was evaluated.

The auscultation method used as a reference (gold standard) of a non-invasive blood pressure (NIBP) measurement method was used. The first blood pressure measurement was performed once each (reference BP not used for evaluation, R0; test BP not used for evaluation, T0) with auscultation and the test medical device (BM5 equipped with BN1 (BNiBP)). The blood pressure used for evaluation was measured four times by auscultation (first reference BP to fourth reference BP, R1 to R4) and three times by the test medical device (first test BP to third test BP, T1 to T3) alternately. A minimum interval of 1 min was allowed between each blood pressure measurement.

Three data pairs (mean value of R1, R2 & T1 / R2, mean value of R3 & T2 / R3, mean value of R4 & T3) were obtained from one study subject. This study aims to verify that the mean value of the differences and standard deviations of data pairs meet the criteria of ISO 81060-2:2018.

ELIGIBILITY:
Inclusion Criteria:

* Recruitment is made through the recruitment notice for patients and their guardians who visit Hanyang University Hospital. Subjects who meet the criteria presented in ISO 81060-2:2018 Protocol 5.1 Subject requirements are recruited.

Exclusion Criteria:

* Emergency surgery patient
* Persons who have mental disorders such as mental retardation, autism, etc. and who have difficulty measuring blood pressure or are expected to have difficulties
* A person who disagreed with the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hoon-Ki Park, M.D., Ph.D., Principal Investigator — Department of Family Medicine, Hanyang University Seoul Hospital
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alpert BS. Validation of the Welch Allyn Spot Vital Signs blood pressure device according to the ANSI/AAMI SP10: 2002. Accuracy and cost-efficiency successfully combined. Blood Press Monit. 2007 Oct;12(5):345-7. doi: 10.1097/MBP.0b013e3282c9abf7. PMID 17890975
- [Background] Coleman A, Freeman P, Steel S, Shennan A. Validation of the Omron 705IT (HEM-759-E) oscillometric blood pressure monitoring device according to the British Hypertension Society protocol. Blood Press Monit. 2006 Feb;11(1):27-32. doi: 10.1097/01.mbp.0000189788.05736.5f. PMID 16410738
- [Background] Guidelines for Accuracy Evaluation of Electronic Sphygmomanometers - KFDA Food and Drug Administration
- [Background] O'Brien E, Atkins N, Stergiou G, Karpettas N, Parati G, Asmar R, Imai Y, Wang J, Mengden T, Shennan A; Working Group on Blood Pressure Monitoring of the European Society of Hypertension. European Society of Hypertension International Protocol revision 2010 for the validation of blood pressure measuring devices in adults. Blood Press Monit. 2010 Feb;15(1):23-38. doi: 10.1097/MBP.0b013e3283360e98. No abstract available. PMID 20110786
- [Background] Stergiou GS, Alpert B, Mieke S, Asmar R, Atkins N, Eckert S, Frick G, Friedman B, Grassl T, Ichikawa T, Ioannidis JP, Lacy P, McManus R, Murray A, Myers M, Palatini P, Parati G, Quinn D, Sarkis J, Shennan A, Usuda T, Wang J, Wu CO, O'Brien E. A universal standard for the validation of blood pressure measuring devices: Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) Collaboration Statement. J Hypertens. 2018 Mar;36(3):472-478. doi: 10.1097/HJH.0000000000001634. PMID 29384983
- [Background] International Organization for Standardization. Noninvasive sphygmomanometers: part 2: clinical investigation of intermittent automated measurement type. (2018): 36.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is made through the recruitment notice for patients and their guardians who visit Hanyang University Hospital. Subjects who meet the criteria presented in ISO 81060-2:2018 Protocol 5.1 Subject requirements are recruited.
Pre-assignment Details: [Selection Criteria] - Subjects who have consented to participate in the clinical trial and voluntarily consented in writing - Subjects who meet the criteria presented in ISO 81060-2:2018 Protocol 5.1 Subject requirements [Items excluded from clinical trials] - Complete blood pressure range recruitment (Range complete) - Arrhythmia - Device failure - Cuff size unavailable - Poor quality of Korotkoff sounds - Observers disagreement - Other factors
Units Other Than Participants: Data pair
Groups:
- Blood Pressure Measurement Group: In this study, the protocol applied to automatic electronic blood pressure system module BN1 for performance evaluation is ISO's proposed "ISO 81060-2:2018 Non-invasive sphygmomanometers- Part2: Clinical investment of internal automatic measurement type". The initial BP measurement is performed alternately, measuring the blood pressure by the measurer and the test device once each, and measuring blood pressure by the measurer four times by the observer and three times by the test device.
  A total of 86 study subjects were enrolled. Three data pairs (mean value of R1, R2 & T1 / R2, mean value of R3 & T2 / R3, mean value of R4 & T3) were obtained from one study subject, and a total of 258 data pairs were obtained. Among them, some data of three study subjects did not satisfy the conditions required by ISO 81060-2:2018, so one dropout data pair (total of three dropout data pairs) occurred. Therefore, 255 valid data pairs were obtained from 86 study subjects.
Period: Overall Study
Arm/Group | Blood Pressure Measurement Group
Started | 86; 258 Data pair
Completed | 86; 255 Data pair (Among them, some data of three study subjects did not satisfy the conditions required by ISO 81060-2:2018, so one dropout data pair (total of three dropout data pairs) occurred. Therefore, 255 valid data pairs were obtained from 86 study subjects.)
Not Completed | 0; 3 Data pair

BASELINE CHARACTERISTICS:
Arm/Group | Blood Pressure Measurement Group
Number analyzed (Participants) | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41
  Between 18 and 65 years | 44
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (18.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 49
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 86

OUTCOME MEASURES:

1. Primary Outcome: Test Device's Blood Pressure of Resting Condition
Description: The blood pressure used for evaluation was measured four times by auscultation (first reference BP to fourth reference BP, R1 to R4) and three times by the test medical device (first test BP to third test BP, T1 to T3) alternately. A minimum interval of 1 min was allowed between each BP measurement. Three data pairs (mean value of R1, R2 & T1 / R2, mean value of R3 & T2 / R3, mean value of R4 & T3) were obtained from one study subject.
  Criterion 1 is that for valid data pairs, the mean value of the difference between the test medical device and the auscultation method BP (test device BP - auscultation BP) should be 5 mmHg or less and the standard deviation (SD) should be 8 mmHg or less.
  Criterion 2 is that, for study subjects, the ISO 81060-2:2018 for presenting different SD thresholds depending on the mean value of the difference should be satisfied. When mean value of the difference is ±1.6, ±0.0 mmHg, the SD should be less than 6.76 and 6.95 mmHg, respectively.
Time Frame: Right after the experiment
Population: A total of 86 study subjects were enrolled. Three data pairs (mean value of R1, R2 & T1 / R2, mean value of R3 & T2 / R3, mean value of R4 & T3) were obtained from one study subject, and a total of 258 data pairs were obtained. Among them, some data of three study subjects did not satisfy the conditions required by ISO 81060-2:2018, so one dropout data pair (total of three dropout data pairs) occurred. Therefore, 255 valid data pairs were obtained from 86 study subjects.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: Data pair
Arm/Group | Blood Pressure Measurement Group
Number analyzed (Participants) | 86
Number analyzed (Data pair) | 255
mmHg
  Criterion 1 (SBP) | -1.55 (6.25)
  Criterion 1 (DBP) | -0.02 (6.61)
  Criterion 2 (SBP) | -1.6 (4.97)
  Criterion 2 (DBP) | -0.0 (5.82)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Blood Pressure Measurement Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT06609486/Prot_SAP_000.pdf